CLINICAL TRIAL: NCT06229561
Title: Soft Tissue Graft Versus Acellular Dermal Matrix in Preservation of Buccal Plate of Bone After Immediate Implant Placement
Brief Title: Soft Tissue Graft Versus Acellular Dermal Matrix in Preservation of Buccal Plate of Bone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Nehal Mohamed Ibrahim Abbas, Principle investor, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nmohamed
Record Dates: First submitted 2023-12-29; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Comparative Study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADM and SCTG (Experimental): ADM and SCTG
  Interventions: Combination Product: Acellular Dermal Matrix
- Acellular Dermal Matrix and soft tissue graft (Experimental): 12participatent in two groups
  Interventions: Combination Product: Acellular Dermal Matrix

INTERVENTIONS:
Combination Product: Acellular Dermal Matrix — Feasibility of soft tissue graft after immediate implant placement

SUMMARY:
Comparative study between 2 groups to assess the feasibility of using Acellular dermal matrix vs Soft tissue Graft after immediate implant placement

DETAILED DESCRIPTION:
It was conclude that SCTG is the gold standard for soft tissue augmentation up till now, However ADM can be alternative to autogenous soft tissue graft.

ELIGIBILITY:
Inclusion Criteria:

Medically free

Exclusion Criteria:

Heavy smoking

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Buccal bone thickness | 6 months follow up
  Assess the buccal bone thickness before and after the graft application

CONTACTS AND LOCATIONS:
Overall Officials: Azhar Journal, Principal Investigator — No affliction
Locations (1):
- Azhar University, Nāşir, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Soft tissue graft versus acellular dermal matrix in preservation of buccal plate of bone after immediate implant placement
Supporting Information: Study Protocol
Time Frame: 6 months follow up
Access Criteria: https://www2.cloud.editorialmanager.com/azjd/default2.aspx
URL: http://www2.cloud.editorialmanager.com/azjd/default2.aspx

REFERENCES:
- [Result] Elaskary A, Abdelrahman H, Elfahl B, Elsabagh H, El-Kimary G, Ghallab NA. Immediate Implant Placement in Intact Fresh Extraction Sockets Using Vestibular Socket Therapy Versus Partial Extraction Therapy in the Esthetic Zone: A Randomized Clinical Trial. Int J Oral Maxillofac Implants. 2023 May, Jun;38(3):468-478. doi: 10.11607/jomi.9973. PMID 37279214